CLINICAL TRIAL: NCT00698698
Title: Tear Proteins and Diabetic Retinopathy
Brief Title: Study on Tear Proteins in Diabetic Retinopathy of Type 2 Diabetics
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Dr.Jamshed Ahmed Assistant Professor, Dow university of Health Sciences Karachi Pakistan
Other Study IDs: Tear proteins
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus
Keywords: tear proteins; diabetic retinopathy; HPLC; Mass spectroscopy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Non diabetic: Normal age and sex matched population
- Grade 1: Diabetic population with no retinopathy or Mild non proliferative diabetic retinopathy
- Grade 2: Moderate non proliferative diabetic retinopathy
- Grade 3: Severe non proliferative diabetic retinopathy
- Grade 4: Proliferative diabetic retinopathy and advanced diabetic eye disease

SUMMARY:
Diabetes mellitus is becoming a global epidemic. There is a need to devise a non invasive method for detection of diabetes and its related complication. Tear proteins are easy to collect causing no harm to a patient and different studies indicate that tear proteins of diabetic patients are significantly different from non diabetic population. This difference in the composition of tear proteins become more pronounced with advancement of diabetic retinopathy.

DETAILED DESCRIPTION:
Diabetes mellitus causes a significant alteration in tear proteins. If we analyze tear proteins by means of electrophoresis, HPLC, and mass spectroscopy.

We can find different type of tear proteins in different grades of diabetic retinopathy these biomarkers can help in mass screening , diagnosis and management of diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with type 2 diabetes
* age above 30
* willing to participate

Exclusion Criteria:

* ocular surface disorders.
* collagen vascular diseases
* Limbal hyperemia
* previous ocular surgery
* creatinine level above 1.0
* liver diseases

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic population
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jamshed Ahmed, FCPS, Principal Investigator — Dow University of Health Sciences Pakistan
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan